

Helicobacter Pylori Eradication Therapy in Portugal: Prospective, randomized, blind and multicentre trial on the efficacy of quadruple therapies and their clinical impact, and immunological and gut microbiota changes

# **INFORMED CONSENT**

February 19<sup>th</sup>, 2021



Helicobacter Pylori Eradication Therapy in Portugal: Prospective, randomized, blind and multicentre trial on the efficacy of quadruple therapies and their clinical impact, and immunological and gut microbiota changes

Gastroenterology Department, Centro Hospitalar e Universitário de Coimbra, E.P.E., Coimbra, Portugal

# INFORMATION FORM AND INFORMED CONSENT

#### **TITLE OF THE RESEARCH PROJECT:**

Helicobacter Pylori Eradication Therapy in Portugal: Prospective, randomized, blind and multicentre trial on the efficacy of quadruple therapies and their clinical impact, and immunological and gut microbiota changes

STUDY PROMOTER: Prof. Dr. Nuno Almeida

RESEARCH COORDINATOR Nuno Almeida

**STUDY CENTRE** Serviço de Gastrenterologia do CHUC

PRINCIPAL INVESTIGATORS Elisa Gravito-Soares, Marta Gravito-Soares

ADRESS Praceta Prof. Mota Pinto, 3000-075 Coimbra

**PHONE NUMBER** (+351)239400483

**FAX NUMBER** (+351)239701517

# **PATIENT'S NAME** (Press letter)

Participants are voluntarily invited to be included in this study, in which will be necessary to take blood and stool samples before and after Helicobacter pylori (Hp) eradication therapy to study the intestinal flora and immunological profile. This procedure, so-called **informed consent**, describes the purpose of the study, the procedures to be performed and the possible benefits and associated risks. The participation of the patient may contribute to improve the knowledge and optimize the therapy of gastric Hp infection.

Participants will receive a copy of this Informed consent to review and seek advice from family and friends (if desired). Investigators and other members of research team will clarify any questions about the consent form. Once the study is understood and there is no doubt about it, the participant should make the decision to participate or not. If the patient agrees to participate, he/she will be asked to sign and date this form. After the participant and investigator's signatures have been obtained, a **copy** of signed informed consent will be given to the participant. In case of no participation, there will be no penalty for the health care provided to the patient.



# 1. GENERAL INFORMATION AND OBJECTIVES OF THE STUDY

This study will take place at the **Gastroenterology Department** of the **Centro Hospitalar e Universitário de Coimbra, E.P.E.** (medical consultation, collection of blood and stool samples) and **Faculties of Medicine and Pharmacy** of the **University of Coimbra** (analysis of gut microbiota in feces and laboratory analysis of blood samples), with the aim of evaluating the influence of different Hp eradication schemes on gut microbiota and immunological profile. This is a multicenter, observational, prospective study, so no changes will be made to your usual medication or treatments other than Hp eradication therapy.

This study was approved by the Ethics Committee of the Faculty of Medicine of the University of Coimbra (FMUC) in order to ensure the rights protection, safety and wellbeing of all included participants and to guarantee public proof of such protection.

In order to ensure participants' safety, the **surveillance** and **support** from a **Gastroenterologist** will be provided before, during and after the Hp eradication therapy.

This study aims to evaluate the influence of Hp eradication therapy on the gut microbiota and its clinical implications including immunological profile, as well as to compare different therapeutic regimens for Hp eradication (all of them currently approved for the treatment of gastric Hp infection).

#### 2. PROCEDURES AND STUDY DESIGN

#### 2.1. Procedures

A Gastroenterologist of the study will conduct a review of medical history and chronic medication from all participants. After the patient accepts to participate in this study, blood and stool samples will be taken before and after Hp eradication therapy. Hp eradication therapy regimens approved for the treatment of gastric Hp infection will be used, including proton pump inhibitors and various antibiotics, for a total duration of 10 to 14 days.

#### 2.2. Schedule of hospital visits and duration

This study consists of 4 gastroenterology medical appointments, lasting about 15 to 20 minutes each, that would already take place for the usual treatment of Hp gastric infection with indication for treatment of the same. In all consultations you will be accompanied by a Gastroenterologist, involving the collection of blood samples in the 1st and 3th/4th consultations, and stool samples in the first 3 consultations. Treatment for Hp eradication will take place between the 1st and 2nd appointments. At the 4th visit, you will also have a breath test to confirm Hp eradication or an upper digestive endoscopy, depending on the clinical indication. If eradication cannot be achieved with the first treatment regimen, you will be directed to alternative eradication therapies.

#### 2.3. Data processing

Data collected from the clinical history and lab results of blood and feces sample analysis will be submitted to a statistical analysis, with anonymity guarantee in all phases of the study.

#### 3. RISKS AND POTENTIAL DRAWBACKS FOR THE PARTICIPANT

The risks of participating in this study are minimal and are the same as for venipuncture for blood collection (pain, bruising, or infection at the puncture site), the same as for blood testing for other purposes. There are no risks associated with stool sampling.

# **4. POTENTIAL BENEFITS**

This study has the advantage of studying gastric infection by Hp and allowing for a better understanding of this disease, its treatment and associated complications. So, this study of Hp eradication therapy and its clinical impact will improve clinical health care offered for patients in similar conditions.

### **5. NEW INFORMATIONS**

Participants will be informed of any new information that may be relevant to Hp gastric infection' condition or influence in their willingness to continue participating in the study.



#### 6. VOLUNTARY PARTICIPATION/ABANDONMENT

Participants are entirely free to accept or refuse to participate in this study, and may withdraw their consent at any time with no any consequence, penalty or loss of benefit and without compromising the relationship between participants and medical team involved in this study. Participants should inform the investigator of their decision to withdraw consent.

Study investigator may decide to end patients' participation, in case of not be in their health best interest to continue in this study. In addition, patients' participation may also be ended in case of no follow the study plan, by administrative decision or decision of the Ethics Committee. Study investigator will notify the participants if one of these conditions is met.

#### 7. CONFIDENTIALITY

Without violating confidentiality rules, auditors and regulatory authorities will be permitted access to medical records to verify the performed procedures and the information obtained from the study in accordance with applicable laws and regulations. Participants' data will be kept confidential and anonymized and in case of study publication, their identity will remain confidential. By signing this informed consent, participants authorize this conditional and restricted access. Participants may also exercise their right to access the information at any time, having access to their medical information directly or through study investigators, and have the right to object to the data transmission that is covered by professional confidentiality.

Identifying medical records and the signed informed consent form will be checked for study purposes by the sponsor and/or representatives of the sponsor, and for regulatory purposes by the sponsor and/or representatives of the sponsor and regulatory agencies in other countries. The Ethics Committee responsible for this study may request access to participants' medical records to ensure that the study is being conducted in accordance with the protocol. Absolute confidentiality cannot be guaranteed due to the need for transmission of information to these parts.

By signing this informed consent form, participants allow that their medical data be verified, processed and reported as necessary for legitimate scientific purposes.

#### Confidentiality and processing of personal data

Personal data of study participants, including medical or health information, collected or created as part of the study (such as medical data or test results), shall be used for carried out the study, including for scientific research related to the condition under study.

In giving consent to participate in this study, the participants' information, including clinical data, shall be used as follows:

- 1. The sponsor, investigators and others involved in the study will collect and use participants' personal data for the purposes described above.
- 2. Study data associated with participants' initials or other code with no direct identification (and no participants' name) will be communicated by researchers and others involved in the study to the study sponsor, who will use them for the purposes described above.
- 3. Study data associated with participants' initials or other code with no direct identification may be communicated to national and international health authorities.
- 4. Participants' identity will not be revealed in any reports or publications resulting from this study.
- 5. All persons or entities with access to participants' personal data are subject to professional confidentiality.
- 6. By giving consent to participate in this study, participants authorize the sponsor or study monitoring companies specifically contracted for this purpose and their employees and/or health authorities, to access the data contained in clinical files, to check the information collected and recorded by the investigators, namely to ensure data accuracy concerning participants and to guarantee that the study is being carried out correctly and the obtained data are reliable.
- 7. Considering law terms, participants have the right, through one of the study investigators, to request access to their data, as well as to request the rectification of their identification data.
- 8. Participants also have the right to withdraw their consent at any time by notifying the investigator, implying the end of participation in the study. However, non-identifiable data collected or created as a part of the study until that time may continue to be used for the purpose of the study, in particular to maintain the scientific integrity of the study, not being removed their medical data from the study file.
- 9. If participants do not give their consent, by signing this document, their participation in this study is not allowed. If and until the given consent is not withdrawn, it remains valid.



# **8. COMPENSATION**

This study is the initiative of the investigator and therefore patient participation is requested without any financial compensation for its implementation, as is also the case with the investigators and the Study Centre.

# 9. CONTACTS

If any questions regarding participants' rights in this study, please contact the Ethics Committee:

The Ethics Committee of the FMUC,

Azinhaga de Santa Comba, Celas – 3000-548 Coimbra

Phone number: (+351)239857707 e-mail: <a href="mailto:comissaoetica@fmed.uc.pt">comissaoetica@fmed.uc.pt</a>

In case of any question about this study, please contact:

Elisa Gravito-Soares, Marta Gravito-Soares

Gastroenterology Department, Centro Hospitalar e Universitário de Coimbra, E.P.E.

Praceta Prof. Mota Pinto, 3000-075 Coimbra, Portugal

Phone number: (+351)239400483



THIS INFORMED CONSENT FORM SHOULD NOT BE SIGNED WITHOUT THE PARTICIPANTS HAVING BEEN GIVEN THE OPPORTUNITY TO ASK AND RECEIVE SATISFACTORY ANSWERS TO ALL THEIR QUESTIONS.

# INFORMED, FREE, AND CLARIFIED CONSENT for participation in Research Study

Please read the following information carefully. If you feel that anything is unclear, please feel free to ask for more information.

<u>Study Title</u>: Impact of Helicobacter pylori eradication therapy on gut microbiota and clinical implications: a prospective observational multicenter randomized blinded study

<u>Background</u>: This clinical research study consists of a national multicenter randomized blinded prospective study, with the purpose of knowing the changes in the gut microbiota induced by different Helicobacter pylori eradication therapy regimens, in order to choose the eradication therapy regimen for Helicobacter pylori that provides the highest efficacy rate and least negative impact on the gut microbiota and consequently the lowest incidence of diseases associated with this change, such as obesity, diabetes mellitus, infectious complications, and autoimmune diseases.

**Explanation of the study**: To carry out this study it is necessary to collect blood and stool samples (before and after Helicobacter pylori eradication therapy) and your authorization to provide your clinical data, which will be deprived of any identification regarding the person in question, which will later be analyzed and published.

<u>Conditions and funding</u>: Your acceptance to participate in this research is voluntary and free of charge, and you will not suffer any prejudice, welfare or other, should you choose not to participate.

<u>Confidentiality and anonymity</u>: The data collected for this study are confidential and anonymity will be assured at all study phases.

I confirm that I have explained to the participant named below the nature, objectives and potential risks of the above Study.

| Researcher: | |
|---|---|
| Name: | |
| Signature: | |
| l, | (Full Name) give my consent for the clinical data |
| concerning my person/relative | (Full Name) (delete as |
| appropriate), regarding the treatment of gastric infection by Helicobacter pylori and changes of the gut microbiota in follow-up in | |
| the Healthcare institution | in Portugal, to be made available for |
| the research study entitled "Helicobacter Pylori eradication Therapy in Portugal: Prospective, randomized, blind and multicentre | |
| trial on the efficacy of quadruple therapies and their clinical impact, and immunological and gut microbiota changes". The | |
| information provided is confidential, ensuring the anonymity of the person concerned. | |
| Participant/Legal Representative: | |
| Signature: | Date: / / |

By signing this document, you declare that you have read and understood this document as well as the verbal information provided to me by the person/s signing above. I have been assured that I may, at any time, refuse to participate in this study without any consequences. Therefore, I agree to participate in this study and allow the use of the clinical data concerning the treatment of gastric infection by Helicobacter pylori and alteration of the intestinal flora, trusting that they will only be used for this research and the guarantees of confidentiality and anonymity given to me by the researcher.



In accordance with the Helsinki Declaration of the World Medical Association and its updates, the participants declare that:

- 1. Read this informed consent form and accept to participate in this study on a voluntary basis.
- 2. Receive all the study information about its nature, objectives, risks, likely duration as well as what is expected from the participant.
- 3. Have the opportunity to ask questions about the study and have understood the answers and the given information.
- 4. At any time can ask further questions to the study investigator and receive information about the study development. The investigator in charge of the study will give to participants all important information that comes up during the study that may change their willingness to continue to participate.
- 5. Agree to use information, including medical history and treatments with strict respect for medical secrecy and anonymity. Participants data will be kept strictly confidential. The authorization for consult their data will be given only to persons designated by the promoter and representatives of regulatory authorities.
- 6. Agree to follow all instructions given during the study and to cooperate with the investigator and to inform him/her immediately of changes in health and well-being and of all unexpected and unusual symptoms that occur.
- 7. Agree to use the results of the study for scientific purposes only and, in particular, I accept that these results will be disclosed to the relevant health authorities.
- 8. Accept that data generated during the study will be computerized by the sponsor or another person designated by him.
- 9. Can exercise their right of rectification and/or opposition.
- 10. Are free to withdraw from the study at any time, without having to justify their decision and without compromising the quality of health care provided. In addition, the investigator has the right to decide on their early withdrawal from the study, with information to the participants about the withdrawal cause.
- 11. Have been informed that the study may be interrupted by decision of the investigator, sponsor or regulatory authorities.

THIS DOCUMENT CONSISTS OF 2 PAGES AND IS MADE UP IN DUPLICATE: ONE COPY FOR THE INVESTIGATOR, ONE FOR THE CONSENTING PERSON